CLINICAL TRIAL: NCT06389812
Title: Dynamic Neurovascular and Cognitive Response to Dual-task Exercise in People With Cognitive Impairment
Brief Title: Dual-task Exercise in People With Cognitive Impairment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Ahmet Begde, Research Associate, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LoughboroughUni
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Dementia; Mild Cognitive Impairment; Older Adults
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual-task group (Experimental): . The motor-cognitive dual-task group will be additionally asked to do horizontal eye movements by watching a TV screen and following a duck moving from side to side (bilateral condition) while performing strengthening exercises. only one session 30 mins.
  Interventions: Other: Dual-task exercise traning
- eye movement exercise group (Active Comparator): asked to do horizontal eye movements by watching a TV screen and following a duck moving from side to side (bilateral condition) while performing strengthening exercises. The duck moves successively between left and right banks of a river at a rate of 500 ms (Brunyé et al., 2009) which was previously found to improve cognitive function. only one session 30 mins.
  Interventions: Other: Dual-task exercise traning
- control (No Intervention): listening a podcast. only one session 30 mins.

INTERVENTIONS:
Other: Dual-task exercise traning — To assess the dynamic effects of each intervention, only one session (30 mins) will be provided. The chair-based exercise session consists of three parts 5 min of active stretching exercises to warm-up, 20 mins of resistance band exercises in a sitting position (Elliott-King et al., 2019) (please see the link for detailed descriptions for seated resistance band workout) and 5 min of passive stretching exercises to cold down. The motor-cognitive dual-task group will be additionally asked to do horizontal eye movements by watching a TV screen and following a duck moving from side to side (bilateral condition) while performing strengthening exercises. The duck moves successively between left and right banks of a river at a rate of 500 ms (Brunyé et al., 2009) which was previously found to improve cognitive function
  Arms: Dual-task group; eye movement exercise group

SUMMARY:
The purpose of this study is to explore how performing two exercise-based tasks simultaneously (dual-task exercise) affects the neurovascular and cognitive responses of people with cognitive impairment, which is a growing concern globally. Specifically, the study will examine how motor-cognitive dual-task exercises, such as using elastic resistance bands combined with visual perception training, including eye movement exercises, can immediately improve outcomes such as Brain-derived neurotrophic factor (BDNF) levels, cerebral blood flow, cognitive function, and mobility. BDNF is a special chemical in our brain that helps with the connections between brain cells. Participants will be asked to complete a single 30-minute exercise session and undergo assessments before and after the intervention. Participants with cognitive impairment will be initially assessed using Mini-Mental State Examination (MMSE) which is a 30-point questionnaire used extensively in clinical and research settings to measure cognitive impairment. Any score of 24 or more (out of 30) indicates normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points), or mild (19-23 points) cognitive impairment. Participants with lower MMSE scores (<10) will be removed from the study.

ELIGIBILITY:
Inclusion Criteria:

* Age >65 (PwD or cognitively impaired older adults) (ICD-10)
* People with and without cognitive impairment (MMSE score 13-30)
* Subjects must be able to exercise at a moderate intensity level (see exclusion criteria)
* Subject must be willing and able to provide a blood sample

Exclusion Criteria:

* • Subjects with other neurological disease (stroke, Parkinson's, or multiple sclerosis)

  * Significant current orthopaedic (fractures, hemiplegia, pain, arthritis etc.), cardiovascular and pulmonary conditions (arrhythmias, uncontrolled hypertension, acute bronchitis, cardiac insufficiency etc.) that would limit the ability to perform cardio-respiratory fitness assessment, tasks or exercise
  * Psychiatric conditions (depression, anxiety disorder, etc.) and a history of severe psychiatric disorders (schizoaffective/bipolar disorders, or schizophrenia)
  * Severe vision/hearing impairments that cannot be corrected with aids
  * Unable to comprehend questionnaire material study procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
BDNF serum level | before and immediately after treatment
  Blood samples will be drawn from the antecubital vein by venepuncture in dry vacuum tubes immediately before the beginning of the exercise training and within 5 min from the termination of the exercise session. Serum will be obtained by the centrifugation of blood (2,000 g for 10 min, 4°C) and then all serum samples will be stored at -80°C until analysis (Máderová et al., 2019).

SECONDARY OUTCOMES:
Visual screening | before and immediately after treatment
  visual processing speed

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided